CLINICAL TRIAL: NCT04806620
Title: Unhide® Project Also Known as The Unhide® Solve Together Unified Platform
Brief Title: Unhide® Project: A Digital Health Platform to Collect Lifestyle Data for Brain Inflammation Research
Status: Recruiting | Type: Observational
Sponsor: Brain Inflammation Collaborative (Other)
Collaborators: Solve ME/CFS Initiative (Other); Care Evolution (Unknown); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19 Syndrome; ME/CFS; Rheumatic Arthritis; Juvenile Rheumatoid Arthritis (JRA); Psoriatic Arthritis (PsA); Ankylosing Spondylitis (AS); Autoimmune Encephalitis; Celiac Disease; Celiac Disease in Children; Chronic Lyme Disease; Post-treatment Lyme Disease Syndrome; Crohn's Disease; Dysautonomia; Anorexia Nervosa; Bulimia Nervosa; ARFID; Avoidant / Restrictive Food Intake Disorder; Ehlers Danlos Syndrome; Endometriosis; Fibromyalgia (FM); Long COVID; Lupus; Migraines; Mast Cell Activation Syndrome; Multiple Sclerosis; Myalgic Encephalomyelitis (ME); Myasthenia Gravis, Generalized; Myasthenia Gravis in Children; Narcolepsy; Obsessive Compulsive Disorder (OCD); PANDAS; Pediatric Acute-onset Neuropsychiatric Syndrome (PANS); POTS - Postural Orthostatic Tachycardia Syndrome; General Anxiety Disorder, Social Anxiety Disorder; PTSD - Post Traumatic Stress Disorder; Psoriasis; Traumatic Brain Injury; Tourette's Syndrome; Inflammatory Bowel Disease (IBD); Autoimmune Diseases; Neurological Diseases or Conditions; Psychiatric Disorder; Sjogren's Syndrome; Ulcerative Colitis and Crohn's Disease
Keywords: Long COVID; Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; Longitudinal Natural History Study; Observational; Neuroinflammatory Disease; Brain inflammation; Neuroinflammatory disorders; PANS/PANDAS; Autoimmune encephalitis; ME/CFS; Dysautonomia / POTS; Multiple sclerosis; Autoimmune disease; Inflammatory bowel disease (Crohn's, ulcerative colitis); Celiac disease; Migraines; Mood disorders (anxiety, depression, bipolar, PTSD, OCD); Mobile health app; Patient registry; Wearable devices; Fatigue; Post-exertional malaise; Brain Fog; Mental health
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic; Rheumatic Fever; Arthritis, Juvenile; Arthritis, Psoriatic; Spondylitis, Ankylosing; Autoimmune Diseases of the Nervous System; Celiac Disease; Post-Lyme Disease Syndrome; Crohn Disease; Autonomic Nervous System Diseases; Anorexia Nervosa; Bulimia Nervosa; Avoidant Restrictive Food Intake Disorder; Ehlers-Danlos Syndrome; Endometriosis; Fibromyalgia; Migraine Disorders; Mast Cell Activation Syndrome; Multiple Sclerosis; Myasthenia Gravis; Narcolepsy; Obsessive-Compulsive Disorder; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Pediatric acute-onset neuropsychiatric syndrome; Postural Orthostatic Tachycardia Syndrome; Generalized Anxiety Disorder; Phobia, Social; Combat Disorders; Psoriasis; Brain Injuries, Traumatic; Tourette Syndrome; Inflammatory Bowel Diseases; Autoimmune Diseases; Mental Disorders; Colitis, Ulcerative; Neuroinflammatory Diseases; Encephalitis; Mood Disorders; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Fatigue; Mental Fatigue; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with brain inflammation and related neuroinflammatory conditions: No intervention will be administered.
- Healthy Controls: No intervention will be administered.

SUMMARY:
The unhide® Project is a non-interventional, longitudinal research study designed to establish a secure data repository of demographic, health, and lifestyle information from individuals with brain inflammation and related neuroinflammatory conditions. Participants in the United States aged 2 years and older will provide self-reported health data, biometrics, and symptom diaries through the MyDataHelps™ app (branded as unhide® for this study). The goal is to create comprehensive longitudinal profiles to facilitate research into disease subtypes, causes, diagnostics, and potential treatments, as well as to identify potential participants for future optional studies. "Healthy" individuals without brain inflammation are also eligible to participate.

The digital health research platform used in this study was originally developed and designed by Solve M.E and was called SolveTogether. The Brain Inflammation Collaborative (BIC) expanded upon Solve M.E.'s work to include related diagnoses, pediatric participants, enhance symptom tracking, and more. BIC and Solve M.E. combined Solve Together and unhide®, to create The unhide® Solve Together Unified Platform in 2025.

DETAILED DESCRIPTION:
The unhide® Project is sponsored by the Brain Inflammation Collaborative (BIC), a nonprofit organization dedicated to advancing understanding, diagnosis, and treatment of neuroinflammatory illness. This study will create a secure, long-term repository of demographic, health, lifestyle, biometric, and symptom data from individuals in the United States with brain inflammation and related conditions, as well as unaffected individuals. Data will be collected remotely through MyDataHelps™ by Care Evolution (rebranded as unhide®), a secure mobile and web-based platform enabling eConsent, survey completion, health record linkage, and optional symptom/activity tracking.

Eligible participants are U.S. residents aged 2 years and older, including both self-identified and physician-diagnosed individuals with infection-associated, autoimmune, neuroimmune, inflammatory gastrointestinal, and behavioral/mood disorders, as well as "healthy" individuals. There are minimal exclusion criteria: individuals living outside the U.S., wards of the state, and those with decisional impairment are ineligible. Pregnant women may participate, and prior or concurrent participation in other research studies is permitted.

The study will follow participants for 10 or more years, collecting self-reported health information, comorbidities, medical history, biometrics (e.g., heart rate, sleep, activity), and symptom data to generate comprehensive longitudinal health profiles. This data resource aims to accelerate translational research, identify disease subtypes, uncover causes and risk factors, support the development of diagnostic tests and treatments, and improve outcomes for individuals affected by neuroinflammation.

ELIGIBILITY:
Participants may be either self-diagnosed, or diagnosed by a physician with the following conditions:

* Infection-associated chronic conditions such as Long COVID, chronic Lyme, myalgic encephalomyelitis (ME/CFS), and post-acute neuropsychiatric syndrome (PANS/PANDAS).
* Neuroimmune, developmental, autonomic, and neurological conditions like migraines, dysautonomia, POTS, multiple sclerosis, and autism spectrum disorder.
* Autoimmune diseases such as Lupus, Sjogren's Disease, rheumatoid arthritis, myasthenia gravis, ankylosing spondylitis, and related autoimmune conditions.

Inflammatory gastrointestinal conditions such as Crohn's Disease, Celiac Disease, and ulcerative colitis.

* Behavioral and mood disorders such as anxiety, depression, bipolar disorder, PTSD, eating disorders, OCD, and other related conditions.
* "Healthy" people (without brain inflammation), including unaffected individuals, unaffected individuals in the same household, and unaffected individuals who are married to relatives and family members.
* Have consistent internet access and a cell phone, tablet, or PC since this is an online or app-based platform that requires entering data and completing surveys.
* Currently live in the United States
* Be able to participate in English (stay tuned for updates about the Spanish language version)
* Be willing to share symptom and health data through the platform

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a study of individuals with brain inflammation and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Phenotypic data collection | From Baseline through up to 10 years, with assessments approximately every 4-12 weeks
  Collect, collate, clean, and analyze a large, well-characterized longitudinal dataset to investigate causes, disease progression, and potential treatments for complex chronic conditions, including infection-associated chronic diseases such as ME/CFS, Long COVID, PANS/PANDAS, autoimmune diseases, and neuroimmune disorders characterized at least in part by symptoms of neuroinflammation, including fatigue, brain fog, mood and behavioral changes, or other central or peripheral neurological symptoms.
Subtyping | From Baseline through up to 10 years, with assessments approximately every 4-12 weeks
  Use the patient reported outcomes to identify brain inflammation and other neuroinflammatory disease subtypes.
  * DePaul Symptom Questionnaire - Short Form (DSQ-SF): A survey measuring frequency and severity of symptoms common in ME/CFS and related conditions. Collected at baseline and quarterly thereafter.
  * COMPASS-31:A 31-item questionnaire survey autonomic symptoms including orthostatic intolerance, gastrointestinal, and vasomotor symptoms. Collected starting 1 month after baseline, every 6 months thereafter.
  * Beighton Questionnaire: A quick screening tool for generalized joint hypermobility, assessing flexibility. Collected starting 1 month after baseline, every 6 months thereafter.
Passive data collection | From Baseline through up to 10 years, with assessments approximately every 4-12 weeks
  Collect data from wearables that allow us to track step counts, heart rate variability and other indicators without the burden of participant data entry.

SECONDARY OUTCOMES:
Demographics | From Baseline through up to 10 years, with assessments approximately every 52 weeks
  Record basic demographic information of our Registry population including: age, race, ethnicity, income, education, employment, marital status.
Comorbitities | From Baseline through up to 10 years, with assessments approximately every 4-12 weeks
  Catalog common comorbidities in our registry population. Participants provide information on diagnosed conditions, age of onset, and whether the condition is still active. Their conditions list can be updated over time.
  * Medical Conditions History: A survey on participants' current and past diagnoses. Collected at baseline and updated every 6 months.
  * Family Health History: A survey on health conditions of biological relatives. Collected starting 1 month after baseline; responses may be updated by participants at any time.
Quality of Life and Functional Status | From Baseline through up to 10 years, with assessments approximately every 4-12 weeks
  Quality of life and daily functioning will be assessed using standardized surveys. These include (but not limited to):
  * Short Form-36 (SF-36): A 36-item survey assessing overall health-related quality of life across eight domains, including physical functioning, pain, vitality, and mental health. Administered at baseline and quarterly thereafter.
  * Self-reported Karnofsky Performance Scale: A scale measuring participants' ability to perform daily activities and independence. Administered 1 month after baseline and annually thereafter.
  * FUNCAP-27 (Functional Capacity): A 27-item survey evaluating functional capacity in daily tasks and physical activities relevant to patient well-being. Administered 1 month after baseline and quarterly thereafter.
Symptoms | From Baseline through up to 10 years, with assessments approximately every 4-12 weeks
  We aim to catalogue the common symptoms of brain inflammation and analyze the data for symptom-based phenotypes. We administer surveys to assess the frequency and severity of symptoms (including neuroinflammatory, behavioral, fatigue, etc.) over time and provide access to a mobile app so participants can log data on their symptoms as often as daily.
  * Symptom Log: Collected continuously via mobile application, with optional daily entry.
  * Fatigue Severity Scale (FSS): A 9-item scale assessing the impact and severity of fatigue on daily functioning and quality of life. Collected starting 1 month after baseline, then quarterly.
  * GAD-7: A 7-item survey assessing the severity of generalized anxiety symptoms over the past two weeks. Collected at baseline and quarterly thereafter.
  * Brain Fog Questionnaire: A survey measuring cognitive symptoms such as memory and concentration. Currently in development.

OTHER OUTCOMES:
Electronic Heath Record Linkage | 36 months
  Link EHR data to patient-reported outcomes in order to better identify neuroinflammation and neuroinflammatory conditions.
Clinical Study Participation | 36 months
  Use the Unhide Platform to identify and invite eligible patients and controls to participate in clinical studies with academic, CRO, and pharmaceutical partners.

CONTACTS AND LOCATIONS:
Overall Officials: Megan L Fitzgerald, PhD, Principal Investigator — Brain Inflammation Collaborative
Locations (1):
- Brain Inflammation Collaborative, Delafield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
BIC Research Collaborators selected by the Brain Inflammation Collaborative will have access to data reports and biosamples from registry participants, in keeping with criteria of the specific collaborative investigation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available to BIC Research Collaborators as long as the study remains active, and for a period thereafter to be determined.
Access Criteria: BIC Research Collaborators will be selected based on mutual interest and on BIC's assessment that the Collaborator possesses knowledge, experience, and training that will benefit interpretation of registry data, and proposes a meritorious and feasible research project in line with BIC's research goals.

REFERENCES:
- [Derived] Ramiller A, Mudie K, Seibert E, Whittaker S. The Facilitation of Clinical and Therapeutic Discoveries in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome and Related Diseases: Protocol for the You + ME Registry Research Platform. JMIR Res Protoc. 2022 Aug 10;11(8):e36798. doi: 10.2196/36798. PMID 35816681